CLINICAL TRIAL: NCT01295424
Title: FinnResusci: Epidemiology and Cost-effectiveness of Out-Of-Hospital Cardiac Arrest in Finland
Brief Title: Epidemiology and Cost-effectiveness of Out-Of-Hospital Cardiac Arrest in Finland
Acronym: FINNRESUSCI
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, jouni kurola, Chief Physician, Kuopio University Hospital
Other Study IDs: KUH 5070212
Record Dates: First submitted 2011-02-09; First posted 2011-02-14 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Intensive Care Unit; Emergency Medical Service
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group study
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study, no interventions

SUMMARY:
Observational study of all out-of-hospital cardiac arrest during 6 months in regional areas of Helsinki University Hospital and Kuopio University Hospital from activation of EMS system until follow up to 6 months of survival.Simultaneous observation of out-of-hospital cardiac arrest primary survivors admitted to all Finnish ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest patients

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Out-of-hospital cardiac arrest patients
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Actual)
Dates: Start 2010-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Alive at hospital discharge (time frame: Hospital discharge day) | 12 hours
  alive at hospital discharge

SECONDARY OUTCOMES:
CPC (time frame: 1 year after cardiac arrest) | 1 year
  Neurologic outcome (Cerebral Performance Category) at one year after out of hospital cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Silfvast, MD, PhD, Study Director — Helsinki University Central Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland